CLINICAL TRIAL: NCT02922959
Title: A Tailored, Peer-delivered Intervention to Reduce Recurring Opioid Overdoses
Acronym: TTIP-PRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Theresa Winhusen, PhD, Professor; Associate Vice Chair and Division Director of Addiction Sciences, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016-6635; R34DA040862 (NIH)
Record Dates: First submitted 2016-09-30; First posted 2016-10-04 (Estimated); Results first posted 2020-06-24 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Drug Overdose; Opioid-Related Disorders; Drug Addiction; Drug Abuse; Substance Abuse
Keywords: Opioid Substitution Treatment; Telephone intervention; secondary prevention; naloxone
MeSH Terms: conditions — Drug Overdose; Opioid-Related Disorders; Substance-Related Disorders | interventions — Naloxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PTOEND (Active Comparator): PTOEND: Personally-tailored opioid overdose prevention education and naloxone distribution.
  Participants in this arm will be given a NARCAN (naloxone) nasal spray kit and personally-tailored information packet about opioid overdose and treatment.
  Interventions: Drug: naloxone nasal spray kit; Behavioral: Personally-tailored opioid overdose prevention education (information packet)
- PTOEND+PI (Experimental): PTOEND+PI: Personally-tailored opioid overdose prevention education and naloxone distribution, plus Peer Intervention.
  In addition to a NARCAN (naloxone) nasal spray kit and personally-tailored information packet about opioid overdose and treatment, participants randomized to this arm will also receive the experimental Peer Intervention.
  Interventions: Behavioral: Peer Intervention; Drug: naloxone nasal spray kit; Behavioral: Personally-tailored opioid overdose prevention education (information packet)

INTERVENTIONS:
Behavioral: Peer Intervention — The Peer Intervention is a 20-minute telephone call delivered by a Peer Interventionist, who is trained to answer questions about the content of the personally-tailored information packets. The primary goal of the call is for the participant and the Peer Interventionist to have an open exchange of information about medication-assisted treatment (MAT) for opioid use disorder.
  Arms: PTOEND+PI
Drug: naloxone nasal spray kit — Naloxone nasal spray (NARCAN) is a potentially life-saving medication that can stop or reverse the effects of an opioid overdose. This nasal spray is approved by the FDA for reversing OODs and has a favorable side-effects profile. A take-home kit will be provided to the patient participants, which may be useful in the event of a future opioid overdose.
  Other Names: NARCAN
Behavioral: Personally-tailored opioid overdose prevention education (information packet) — Personally-tailored information packet with three participant-specific reports ("Personal Overdose Risk Factors Report"; "Medication Assisted Treatment (MAT) Report"; and the "Opioid Overdose Information Report"), and general written information about opioid overdose and treatment for opioid use disorder.

SUMMARY:
This project will further develop and test the Tailored Telephone Intervention delivered by Peers to Prevent Recurring Opioid Overdoses (TTIP-PRO), a promising, low-cost, intervention to facilitate entry into medication assisted treatment (MAT) for individuals experiencing a non-fatal opioid overdoses (OOD). A prior small-scale pilot/feasibility study of TTIP-PRO (NCT02282306) found that the participating patients and the Peer Interventionists were satisfied with their participation, the intervention was acceptable, and the system for generating patient-tailored intervention information performed well. The overall goal of the present study is to conduct a pilot randomized controlled trial of TTIP-PRO versus a control group. It is hypothesized that patients in the TTIP-PRO group will have more favorable drug-abuse-related outcomes than patients in the control group.

DETAILED DESCRIPTION:
This pilot study is a randomized controlled intent-to-treat (ITT) clinical trial. Approximately eighty eligible participants will be randomized in a 1:1 ratio to the control condition (Information and NARCAN® (naloxone) Nasal Spray kit) or to the experimental condition (TTIP-PRO in addition to the elements provided in the control condition). All participants will complete a follow-up phone call approximately 3-weeks post-randomization, during which process measures will be completed, and in-person visits at approximately 3, 6-, and 12-months following enrollment.

This is a single site study; all data will be collected at the University of Cincinnati. Approximately 80 participants will be randomized into this pilot efficacy trial. The hypotheses to be tested include that participants assigned to the TTIP-PRO intervention will: have a higher rate of enrollment in MAT, have a lower rate of recurring opioid overdose, and have greater reduction in illicit opioid use.

ELIGIBILITY:
Inclusion Criteria:

* Report having been treated for an OOD within the past 6 months
* Age 18 years or older;
* Scores "high risk" for heroin and/or non-medical use of prescription opioids on the National Institute on Drug Abuse modified Alcohol, Smoking and Substance Involvement Screening Test (NIDA-modified ASSIST) (i.e., ≥ 27)
* Be able to understand the study, and having understood, provide written informed consent in English
* Access to a phone (for TTIP-PRO intervention and phone follow-up)
* Be willing to have their intervention audio recorded and rated if randomized to TTIP-PRO
* Have an opioid-positive baseline/screening urine drug screen.

Exclusion Criteria:

* In the judgment of the investigator, would not be expected to complete the study protocol (e.g., due to relocation from the clinic area, probable incarceration, etc.)
* Current engagement in addiction treatment
* Residence more than 40 miles from the location of follow-up visits
* Inability to provide sufficient contact information (must provide at least 2 reliable locators)
* Prior participation in the current study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Winhusen, PhD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati Addiction Sciences Division, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared in a timely manner, i.e., no later than the acceptance for publication of the main findings from the final dataset. The dataset will include information about illegal activities (e.g., illicit opioid use, etc.). Thus, in addition to only a de-identified database being shared, we will also require a data sharing agreement. The data sharing agreement will require commitment to: 1) not re-disclose the data; 2) secure the data; 3) use the data for research purposes only; 4) make no attempt to identify individual participants; 5) destroy the data once the planned research activities have been completed; 6) follow all relevant NIH policies.

REFERENCES:
- [Derived] Kropp F, Wilder C, Theobald J, Lewis D, Winhusen TJ. The feasibility and safety of training patients in opioid treatment to serve as peer recovery support service interventionists. Subst Abus. 2022;43(1):527-530. doi: 10.1080/08897077.2021.1949667. Epub 2021 Jul 8. PMID 34236298

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants were recruited through various methods including advertisements, flyers, and word-of-mouth. Greater than 90% of participants were recruited from a syringe exchange program. All participants were given a thorough explanation of the study and signed an informed consent form.
Pre-assignment Details: 116 potential participants were consented and screened, and 80 were randomized to Personally-tailored opioid overdose education and naloxone distribution plus Peer Intervention (PTOEND+PI) (n=40) or PTOEND (n=40).
Groups:
- PTOEND: PTOEND: Personally-tailored opioid overdose prevention education and naloxone distribution.
  Participants in this arm will be given a NARCAN (naloxone) nasal spray kit and personally-tailored information packet about opioid overdose and treatment.
  naloxone nasal spray kit: Naloxone nasal spray (NARCAN) is a potentially life-saving medication that can stop or reverse the effects of an opioid overdose.
  Personally-tailored opioid overdose prevention education (information packet): Personally-tailored information packet with three participant-specific reports and general written information about opioid overdose and treatment for opioid use disorder.
- PTOEND+PI: PTOEND+PI: Personally-tailored opioid overdose prevention education and naloxone distribution, plus Peer Intervention.
  In addition to a NARCAN (naloxone) nasal spray kit and personally-tailored information packet about opioid overdose and treatment, participants randomized to this arm will also receive the experimental Peer Intervention.
  Peer Intervention: The Peer Intervention is a 20-minute telephone call delivered by a Peer Interventionist, who is trained to answer questions about the content of the personally-tailored information packets.
  naloxone nasal spray kit: Naloxone nasal spray (NARCAN) is a potentially life-saving medication that can stop or reverse the effects of an opioid overdose.
  Personally-tailored opioid overdose prevention education (information packet): Personally-tailored information packet with three participant-specific reports and general written information about opioid overdose and treatment for opioid use disorder.
Period: Overall Study
Arm/Group | PTOEND | PTOEND+PI
Started | 40 | 40
3 Weeks | 38 (n=38 (95.0%)) | 36 (n=36 (90.0%))
3 Months | 35 (n=35 (87.5%)) | 31 (n=31 (77.5%))
6 Months | 28 (n=28 (70.0%)) | 30 (n=30 (75.0%))
12 Months | 21 (n=21 (52.5%)) | 23 (n=23 (57.5%))
Completed | 21 | 23
Not Completed | 19 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PTOEND | PTOEND+PI | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.0 (10.3) | 40.3 (12.5) | 39.1 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 14 | 36
  Male | 18 | 26 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 39 | 39 | 78
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 32 | 32 | 64
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Medication-Assisted Treatment Enrollment
Description: whether or not participant enrolled in medication-assisted treatment within the follow-up period
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | PTOEND | PTOEND+PI
Number analyzed (Participants) | 40 | 40
Participants | 7 | 13

2. Secondary Outcome: Opioid Overdose Experience
Description: whether or not participant experienced an opioid overdose within the follow-up period period.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | PTOEND | PTOEND+PI
Number analyzed (Participants) | 40 | 40
Participants | 13 | 5

3. Secondary Outcome: Change in Opioid Use (Timeline Follow-back)
Description: Difference in self-reported opioid use in the prior 28 days, from Baseline to 12-month visit, computed as: (12-month opioid use days - Baseline opioid use days); negative values indicate a reduction in self-reported opioid use days from Baseline to 12-month visit.
Time Frame: at 12-month visit
Population: Analysis could only be done on data provided by participants who attended the 12-month visit
Measure: Mean (Standard Deviation); unit: days
Arm/Group | PTOEND | PTOEND+PI
Number analyzed (Participants) | 21 | 23
days | -10.2 (12.7) | -8.7 (13.6)

4. Secondary Outcome: Change in Opioid Use (Urine Drug Screen)
Description: Number of participants who provided an opioid-negative urine sample, assessed by a rapid urine drug screen system, at the 12-month visit. Results that were positive, but specific to only buprenorphine or methadone, were counted as negative for participants with verified enrollment in medication-assisted treatment. Note that all participants were required to have an opioid-positive urine sample at Baseline, in order to be eligible for the study.
Time Frame: at 12-month visit
Population: Analysis could only be done on samples provided by participants who attended the 12-month visit
Measure: Count of Participants; unit: Participants
Arm/Group | PTOEND | PTOEND+PI
Number analyzed (Participants) | 21 | 23
Participants | 18 | 20

ADVERSE EVENTS:
Time Frame: 12 months. Adverse events were systematically assessed during each research visit.
Description: Serious Adverse Events were defined as an event that results in any of the following outcomes: death, life threatening, requires hospitalization, initial or prolonged, results in disability, congenital anomaly, requires intervention to prevent permanent impairment or damage, or other significant medical event.
  Other (non-Serious) adverse events were defined as suicidal ideation or homicidal ideation.
Arm/Group | PTOEND | PTOEND+PI
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 9/40 | 7/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PTOEND (N=40) | PTOEND+PI (N=40)
Hospitalization for musculoskeletal problem / injury (Musculoskeletal and connective tissue disorders) | 0 | 3
Suicide Attempt (Psychiatric disorders) | 0 | 1
Congenital Anomaly or Birth Defect (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Hospitalization for nervous system disorder (Nervous system disorders) | 1 | 1
Hospitalization for renal disorder (Renal and urinary disorders) | 0 | 1
Hospitalization related to pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 | 1
Hospitalization for infection/abscess (Infections and infestations) | 2 | 1
Hospitalization for psychiatric problem (Psychiatric disorders) | 2 | 0
Hospitalization for respiratory condition (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hospitalization for multiple causes (General disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/59/NCT02922959/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-11-08): https://cdn.clinicaltrials.gov/large-docs/59/NCT02922959/Prot_SAP_001.pdf